CLINICAL TRIAL: NCT00565760
Title: A Double-Blind, Multi-Center Extension Study to Evaluate the Safety and Efficacy of Q8003 in Patients With Acute Moderate to Severe Pain
Brief Title: Extension Study to Evaluate the Safety of Q8003 in Patients With Acute Moderate to Severe Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q8003-010
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Acute Moderate to Severe Pain
Keywords: Acute; Pain
MeSH Terms: conditions — Pain | interventions — MoxDuo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Q8003
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Q8003 — Capsules
  Arms: 1
Drug: Placebo — Capsules
  Arms: 2

SUMMARY:
This is a Phase 3 double-blind, multiple dose safety extension study of Q8003 administered at daily doses up to 36 mg morphine/24 mg oxycodone (Q8003 36mg/24mg) over a treatment period of up to 4 weeks. Patients with acute moderate to severe pain who have completed participation in one of the designated QRxPharma, Inc. acute pain lead-in studies will be eligible for this trial.

DETAILED DESCRIPTION:
The currently designated acute pain lead-in study is Study Q8003-007, which is a safety and efficacy study of Q8003 in the management of post-bunionectomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed participation in one of the designated eligible QRxPharma, Inc. acute pain lead-in studies.
* Patient has a BMI ≤35.
* Patient will anticipate taking the first dose of study medication in this Extension Study no longer than 24 hours after taking the final dose of study medication in the lead-in study.
* Patient is in good health as determined by the Investigator via physical examination at the Extension Study Baseline Visit.
* If female, patient is at least one year post-menopausal (defined as one year without menses), surgically sterile (must be documented), or practicing effective contraception, in the opinion of the Investigator, and be willing to continue to use effective contraception for the duration of participation in the study.
* If female, patient is non-lactating, and if of child-bearing potential, has a negative urine pregnancy test result at Baseline Visit.
* Patient has a pulse-oximetry measurement ≥95%, a respiration rate ≥12 breaths/minute, systolic blood pressure ≥100 mm Hg, and diastolic blood pressure ≥50 mm Hg at the Extension Study Baseline Visit.
* Patient is willing to refrain from driving throughout the duration of participation in the study.

Exclusion Criteria:

* Patient has acute asthma, head injury, elevated intracranial pressure, convulsive states, congestive heart failure (NYHA classification of III or IV), current cardiac arrhythmia, current transient cerebral ischemic attacks, current uncontrolled unstable co-existent systemic disease, serious intercurrent illness, other medical condition, laboratory abnormality, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study.
* Patient has allergy, hypersensitivity, or contraindications to opioids.
* Patient has poorly controlled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >95 mm Hg despite antihypertensive medication) at the Extension Study Baseline Visit.
* Patient is currently taking tramadol or anticipates taking tramadol during the course of the study.
* Patient is currently taking antipsychotic drugs, monoamine oxidase inhibitors, muscle relaxants, or medications for the treatment of depression.
* Patient is currently taking any opioid analgesic other than Q8003 or other opioid study medication, or anticipates taking any opioid analgesic other than Q8003 or other opioid study medication during the course of the study.
* Patient is at high risk of addiction: patient has a history of substance abuse (excluding nicotine or caffeine), a family history of substance abuse, or a history of adverse consequences related to substance abuse including legal issues.
* Patient has a history of drug or alcohol use or dependence that, in the opinion of the Investigator, would interfere with adherence to study requirements.
* Patient has any medical, psychological, cognitive, social and/or legal conditions that could, in the opinion of the Investigator, compromise patient safety or interfere with the ability of the patient to give informed consent and/or comply with all study requirements, including the necessary time commitment.
* Patient has received any investigational medication within 30 days prior to the first dose of study drug in this study other than Q8003 or is scheduled to receive any investigational drug other than Q8003 during the course of this study.
* Patient has previously been admitted to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety: adverse events | Up to 4 weeks with 3 weeks follow-up

SECONDARY OUTCOMES:
Efficacy: difference in pain intensity scores from baseline | Up to 4 weeks with 3 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Warren Stern, Ph.D., Study Director — QRxPharma Inc.
Locations (6):
- United States (6):
  - Advanced Clinical Research Institute, Anaheim, California
  - Chesapeake Research Group, Pasadena, Maryland
  - Advanced Regional Center for Foot and Ankle Care, Altoona, Pennsylvania
  - Scirex Research Center, Houston, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah